CLINICAL TRIAL: NCT05686265
Title: Cerebral Nitrosative/Oxidative Stress in Aneurysmal Subarachnoid Haemorrhage
Acronym: NOX2
Status: Terminated | Type: Observational
Why Stopped: Practical reasons (project coordinator has resigned and started new employment).
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of South Wales (Other)
Responsible Party: Principal Investigator, Anton Lund, Principal Investigator, Rigshospitalet, Denmark
Other Study IDs: H-22073181
Record Dates: First submitted 2023-01-09; First posted 2023-01-17 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: Oxidative Stress; Nitrosative Stress; Nitric Oxide; Acute Brain Injury; Subarachnoid Hemorrhage; Secondary Brain Injury; Neuromonitoring
MeSH Terms: conditions — Subarachnoid Hemorrhage; Brain Injuries | interventions — Oxygen

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (whole blood, serum, plasma, and red blood cells), cerebrospinal fluid, and cerebral microdialysate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with SAH (see eligibility criteria below).
  Interventions: Drug: Oxygen
- Controls: Healthy controls (see eligibility criteria below).
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — Physiological intervention consisting of 1 hour of mild hypoxia (PaO2 9-10 kPa), 1 hour of mild hyperoxia (PaO2 13-14 kPa), and in healthy subjects also 1 hour of an inspired oxygen fraction of 100%.
  Other Names: Hypoxia and hyperoxia

SUMMARY:
Aneurysmal subarachnoid haemorrhage (SAH) carries a high morbidity and mortality, which is in part due to the development of secondary brain injury. The mechanisms behind this remain incompletely understood, but oxidative/nitrosative stress and disturbances in vasoregulatory mechanisms are believed to be involved. The present study aims to characterise the transcerebral exchange of oxidative/nitrosative stress markers and nitric oxide metabolites during the early phase after SAH compared to healthy volunteers, including the influence of induced changes in arteriel oxygen tension.

DETAILED DESCRIPTION:
BACKGROUND:

Aneurysmal subarachnoid haemorrhage (SAH) carries a high morbidity and mortality. This is in large part due to the development of secondary brain injury, including the complication delayed cerebral ischaemia (DCI), which affects 30% of initial survivors. The mechanisms behind secondary brain injury after SAH are incompletely understood.

Nitric oxide (NO) is a potent endogenous vasodilator produced from arginine by the enzyme nitric oxide synthase (NOS), which exists in three isoforms: endothelial, neuronal, and inducible NOS (eNOS, nNOS and iNOS). In conditions of inflammation and oxidative stress, free radicals may react with NO to form peroxynitrite (ONOO-), which is highly reactive and can directly damage biological macromolecules such as lipids and proteins. This phenomenon, i.e. an increased production of reactive nitrogen species potentially leading to cellular damage, is termed nitrosative stress.

It is widely believed that oxidative/nitrosative stress and associated disturbances in the metabolism of NO are involved in the development of secondary brain injury after SAH, but the exact role of these mechanisms remains incompletely understood. While some authors believe that NOS dysfunction and a resultant low NO bioavailability is an important cause of secondary brain injury (and a key mechanism behind DCI), others argue that an overproduction of NO mediated by iNOS is maladaptive response leading to aggravated tissue injury due to nitrosative stress.

The transcerebral (i.e., arterial to jugular venous) exchange of NO metabolites and its interrelationship with oxidative stress has never been studied in patients with SAH. The investigators hypothesise that SAH is associated with an initial reduction in the cerebrovascular bioavailability of NO due to scavenging by free radicals. This could contribute to a vicious cycle, in which a resulting increase in microvascular resistance, cerebral hypoperfusion, and brain tissue hypoxia further increases free radical production and NO depletion, ultimately leading to ischaemic brain injury and poor outcome.

HYPOTHESES:

The present explorative study will characterise the transcerebral exchange of oxidative/nitrosative stress markers and NO metabolites during the early phase after SAH as compared to healthy volunteers. Additionally, it will examine the influence of these disturbances on indices of brain ischemia and metabolic dysfunction as assessed by multimodal neuromonitoring, and the influence of induced changes in arterial oxygen tension (PaO2). The investigators hypothesise that:

1. Patients will have a greater cerebral efflux of oxidative/nitrosative stress markers and a lower cerebrovascular bioavailability of NO compared to healthy controls.
2. SAH patients will exhibit a progressive decrease in the transcerebral release of oxidative/nitrosative stress markers and a corresponding increase in the cerebrovascular bioavailability of NO in the days following ictus.
3. A greater clinical severity of SAH will be associated with a greater transcerebral release of oxidative/nitrosative stress markers and a lower cerebrovascular bioavailability of NO.
4. A lower brain tissue oxygen tension (PbtO2) and a larger burden of brain tissue hypoxia (defined as the percentage of monitoring time with a PbtO2 <20mmHg) will be associated with a greater cerebral efflux of oxidative/nitrosative stress markers and a lower cerebral bioavailability of NO.
5. A greater microdialysate lactate/pyruvate ratio and a larger burden of brain metabolic crisis (defined as the percentage of monitoring time with a lactate/pyruvate ratio >40 and glucose concentration <0,7 mmol/l) will be associated with a greater cerebral efflux of oxidative/nitrosative stress markers and a lower cerebral bioavailability of NO.
6. Induced mild hypoxia will be associated with an increased transcerebral release of markers of oxidative/nitrosative stress and a reduction in the cerebrovascular bioavailability of NO compared to baseline, while induced mild hyperoxia will have the opposite effect.

METHODS:

The study is a prospective physiological study which will include patients with SAH admitted to the Neurointensive Care Unit (NICU) at Rigshospitalet. Patient inclusion will be continued until we have obtained complete data on 20 patients in the interventional substudy (see below), or until the 1st of April 2024, at which point inclusion will be halted and data will be analysed irrespective of the number of included patients. In addition, 12 healthy subjects will be included to serve as a control group.

Practical conduct of the study, patients:

Patients will have an arterial catheter inserted shortly after admission as part of routine care. In addition, as early as possible after closure of the aneurysm, a retrograde internal jugular venous catheter (RJV catheter) will be inserted for sampling of cerebral venous blood. Vital parameters will be monitored according to standard practice in the NICU, and patients will undergo continuous multimodal neuromonitoring of intracranial pressure (ICP), PbtO2, and brain metabolism (cerebral microdialysis). Additionally, jugular bulb blood pressure will be monitored on the RJV-catheter for at least 24 hours in all patients.

During interventions, transcranial Doppler ultrasound (TCD) will be used to determine middle cerebral artery mean flow velocity as a surrogate measure of cerebral blood flow. The study will consist of an observational and an interventional substudy, which are described individually below.

Observational substudy: Paired blood samples (i.e., simultaneous blood samples from the RJV and arterial catheters) will be drawn 1) immediately after placement of the RJV catheter (expected: day 0-2 after admission), 2) during interventions (see below), and 3) shortly before removal of the RJV catheter (expected: day 3-6 after admission). In addition to blood sampling, patients with an existing external ventricular drain will undergo sampling of CSF, and patients with a cerebral microdialysis catheter will undergo sampling of excess microdialysate for explorative purposes.

Interventional substudy: Mild hypo- and hyperoxia will be induced by in a randomised order by changing ventilator settings (the fraction of inspired oxygen), aiming at a PaO2 of 9-10 kPa for mild hypoxia and 13-14 kPa for mild hyperoxia (standard treatment target: 10-12 kPa). Blood samples will be drawn at baseline (normoxia) and after 60 minutes of each intervention (3 paired blood samples in total).

Practical conduct of the study, healthy controls:

Experiments in healthy subjects will be conducted in the NICU. Instrumentation and monitoring is similar to what is described above: an arterial- and RJV catheter will be inserted, and subjects will undergo TCD monitoring as an index of cerebral blood flow in addition to standard cardiorespiratory monitoring.

After instrumentation and a short rest period, a baseline evaluation will be conducted, after which subjects will undergo interventions in a randomised order: Hypo- and hyperoxia will be induced using a tight-fitting mask connected to a non-rebreathing valve, an end-tidal CO2 monitor, and a reservoir supplied through compressed gas cylinders. The fraction of inspired oxygen will be titrated, aiming at a PaO2 of 9-10 kPa for mild hypoxia and 13-14 kPa for mild hyperoxia.. Additionally, healthy subjects will undergo a third intervention where the fraction of inspired oxygen will be increased to 100%. Isocapnia will be ensured by adding CO2 to the inspired air ad hoc. Blood samples will be drawn at baseline (normoxia) and after 60 minutes of mild hypoxia, 60 minutes of mild hyperoxia, and 60 minutes of "severe hyperoxia".

BIOCHEMICAL ANALYSES:

At each sampling time point, a small amount of blood will immediately be analysed for levels of blood gases and acid-base status. The remaining biological samples will be centrifuged, aliquoted, and stored at -80°C until analysis.

Blood samples will be analysed for the following markers of oxidative stress: the ascorbate radical, lipid hydroperoxides, myeloperoxidase, and the antioxidants glutathione, α/γ-tocopherol, α/β-carotene, retinol and lycopene.

The following NO metabolites will be determined: total plasma NO concentration (nitrate (NO3-) + nitrite (NO2-) + S-nitrosothiols (RSNO)) and total red blood cell bound NO (nitrite (NO2-) + nitrosyl haemoglobin (HbNO) + S-nitrosohaemoglobin (HbSNO)). In addition, 3-nitrotyrosine will be determined as a surrogate marker for peroxynitrite.

The following biomarkers of neurovascular unit injury will be determined: S100ß, glial fibrillary acidic protein, neuron-specific enolase, ubiquitin carboxy-terminal hydrolase L1, neurofilament light-chain and total tau.

Additionally, as part of explorative substudies, blood samples from certain patients may be analysed for leukocyte subsets using mass cytometry, as well as markers of endothelial injury (plasma syndecan-1, soluble thrombomodulin, and PECAM-1).

ELIGIBILITY:
Inclusion Criteria (patients):

* Age ≥ 18 years
* Admission to the NICU at Rigshospitalet
* Diagnosis of aneurysmal SAH
* Need for sedation and mechanical ventilation after the aneurysm has been secured
* Initiation of study possible ≤3 days after the ictus
* Closest relatives understand written and spoken Danish or English

Exclusion Criteria (patients):

* Brain death before inclusion
* Expected death within 24 hours
* Failed or conservative treatment of the aneurysm
* Severe acute lung failure with a PaO2/FiO2-ratio ≤16 kPa
* Severe chronic lung failure with habitual long-term oxygen therapy
* Habitual treatment with medication directly affecting NO metabolism (e.g., sildenafil)

Inclusion Criteria (patients):

* Age 40-60 years
* 50/50 sex distribution (6 men and 6 women)
* Healthy (including no prior cerebrovascular disease)
* No regular medication or recreational drug use
* Understands written and spoken Danish or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twenty patients with severe SAH and twelve pseudo-matched healthy controls.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Transcerebral exchange of bioactive NO, patients vs. controls | At baseline
  Transcerebral exchange of bioactive NO (plasma nitrite + S-nitrosothiols) (nM) in patients vs. controls.
Transcerebral exchange of oxidative stress markers, patients vs. controls | At baseline
  Transcerebral exchange of the ascorbate radical (μM) in patients vs. healthy controls.
Transcerebral exchange of nitrosative stress markers, patients vs. controls | At baseline
  Transcerebral exchange of 3-nitrotyrosine (nM) in patients vs. healthy controls.

SECONDARY OUTCOMES:
Transcerebral exchange of nitrosative/oxidative stress markers, effects of hypo-/hyperoxia | Within one week
  Changes in the transcerebral exchange of nitrosative/oxidative stress markers during hypoxia and hyperoxia, respectively, compared to baseline (normoxia) in both patients and controls.
Transcerebral exchange of nitrosative/oxidative stress markers, changes over time | Within one week
  Changes in the transcerebral exchange of nitrosative/oxidative stress markers over time in patients.

OTHER OUTCOMES:
Nitrosative/oxidative stress, relationship to disease severity | At baseline
  Association between disease severity (i.e., WFNS-score) and the transcerebral exchange of nitrosative/oxidative stress markers in patients.
Nitrosative/oxidative stress, relationship to brain oxygenation | Within one week
  Associations between the transcerebral exchange of nitrosative/oxidative stress markers and the occurrence of brain tissue hypoxia (defined a PbtO2 <20mmHg) in patients undergoing PbtO2-monitoring.
Nitrosative/oxidative stress, relationship to brain metabolism | Within one week
  Associations between the transcerebral exchange of nitrosative/oxidative stress markers and brain metabolic crisis (defined as a lactate/pyruvate ratio >40 and glucose concentration ≤0,7 mmol/l) in patients undergoing cerebral microdialysis.
Endotheliopathy, changes over time | Within one week
  Changes in the transcerebral exchange of markers of endotheliopathy: syndecan-1 (ng/ml), soluble thrombomodulin (ng/ml) and platelet and endothelial cell adhesion molecule 1 (PECAM-1, ng/ml).
Immune cell subsets, changes over time | Within one week
  Changes in the transcerebral exchange of immune cell subsets as evaluated using mass cytometry.
Jugular bulb pressure, relationship to intracranial pressure | Within one week
  Association between jugular bulb pressure (mmHg) and intracranial pressure (mmHg) in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Anton Lund, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data from each individual participant will be available after publication of planned manuscripts, with a valid reason, and after signing a data processing agreement.
Supporting Information: Study Protocol
Time Frame: The approved study protocol will be available upon request until publication of the study results.
Access Criteria: Valid reason and contact with author.

REFERENCES:
- [Background] Suarez JI, Tarr RW, Selman WR. Aneurysmal subarachnoid hemorrhage. N Engl J Med. 2006 Jan 26;354(4):387-96. doi: 10.1056/NEJMra052732. No abstract available. PMID 16436770
- [Background] van Gijn J, Kerr RS, Rinkel GJ. Subarachnoid haemorrhage. Lancet. 2007 Jan 27;369(9558):306-18. doi: 10.1016/S0140-6736(07)60153-6. PMID 17258671
- [Background] Macdonald RL. Delayed neurological deterioration after subarachnoid haemorrhage. Nat Rev Neurol. 2014 Jan;10(1):44-58. doi: 10.1038/nrneurol.2013.246. Epub 2013 Dec 10. PMID 24323051
- [Background] Vergouwen MD, Vermeulen M, van Gijn J, Rinkel GJ, Wijdicks EF, Muizelaar JP, Mendelow AD, Juvela S, Yonas H, Terbrugge KG, Macdonald RL, Diringer MN, Broderick JP, Dreier JP, Roos YB. Definition of delayed cerebral ischemia after aneurysmal subarachnoid hemorrhage as an outcome event in clinical trials and observational studies: proposal of a multidisciplinary research group. Stroke. 2010 Oct;41(10):2391-5. doi: 10.1161/STROKEAHA.110.589275. Epub 2010 Aug 26. PMID 20798370
- [Background] Budohoski KP, Guilfoyle M, Helmy A, Huuskonen T, Czosnyka M, Kirollos R, Menon DK, Pickard JD, Kirkpatrick PJ. The pathophysiology and treatment of delayed cerebral ischaemia following subarachnoid haemorrhage. J Neurol Neurosurg Psychiatry. 2014 Dec;85(12):1343-53. doi: 10.1136/jnnp-2014-307711. Epub 2014 May 20. PMID 24847164
- [Background] Pacher P, Beckman JS, Liaudet L. Nitric oxide and peroxynitrite in health and disease. Physiol Rev. 2007 Jan;87(1):315-424. doi: 10.1152/physrev.00029.2006. PMID 17237348
- [Background] Garry PS, Ezra M, Rowland MJ, Westbrook J, Pattinson KT. The role of the nitric oxide pathway in brain injury and its treatment--from bench to bedside. Exp Neurol. 2015 Jan;263:235-43. doi: 10.1016/j.expneurol.2014.10.017. Epub 2014 Oct 29. PMID 25447937
- [Background] Pluta RM. Delayed cerebral vasospasm and nitric oxide: review, new hypothesis, and proposed treatment. Pharmacol Ther. 2005 Jan;105(1):23-56. doi: 10.1016/j.pharmthera.2004.10.002. PMID 15626454
- [Background] Pluta RM. Dysfunction of nitric oxide synthases as a cause and therapeutic target in delayed cerebral vasospasm after SAH. Acta Neurochir Suppl. 2008;104:139-47. doi: 10.1007/978-3-211-75718-5_28. PMID 18456999
- [Background] Sehba FA, Schwartz AY, Chereshnev I, Bederson JB. Acute decrease in cerebral nitric oxide levels after subarachnoid hemorrhage. J Cereb Blood Flow Metab. 2000 Mar;20(3):604-11. doi: 10.1097/00004647-200003000-00018. PMID 10724124
- [Background] Sobey CG, Faraci FM. Subarachnoid haemorrhage: what happens to the cerebral arteries? Clin Exp Pharmacol Physiol. 1998 Nov;25(11):867-76. doi: 10.1111/j.1440-1681.1998.tb02337.x. PMID 9807657
- [Background] Sehba FA, Bederson JB. Nitric oxide in early brain injury after subarachnoid hemorrhage. Acta Neurochir Suppl. 2011;110(Pt 1):99-103. doi: 10.1007/978-3-7091-0353-1_18. PMID 21116923
- [Background] Sehba FA, Chereshnev I, Maayani S, Friedrich V Jr, Bederson JB. Nitric oxide synthase in acute alteration of nitric oxide levels after subarachnoid hemorrhage. Neurosurgery. 2004 Sep;55(3):671-7; discussion 677-8. doi: 10.1227/01.neu.0000134557.82423.b2. PMID 15335435
- [Background] Hino A, Tokuyama Y, Weir B, Takeda J, Yano H, Bell GI, Macdonald RL. Changes in endothelial nitric oxide synthase mRNA during vasospasm after subarachnoid hemorrhage in monkeys. Neurosurgery. 1996 Sep;39(3):562-7; discussion 567-8. doi: 10.1097/00006123-199609000-00026. PMID 8875487
- [Background] Jung CS, Oldfield EH, Harvey-White J, Espey MG, Zimmermann M, Seifert V, Pluta RM. Association of an endogenous inhibitor of nitric oxide synthase with cerebral vasospasm in patients with aneurysmal subarachnoid hemorrhage. J Neurosurg. 2007 Nov;107(5):945-50. doi: 10.3171/JNS-07/11/0945. PMID 17977265
- [Background] Iqbal S, Hayman EG, Hong C, Stokum JA, Kurland DB, Gerzanich V, Simard JM. Inducible nitric oxide synthase (NOS-2) in subarachnoid hemorrhage: Regulatory mechanisms and therapeutic implications. Brain Circ. 2016;2(1):8-19. doi: 10.4103/2394-8108.178541. PMID 27774520
- [Background] Macmillan CS, Andrews PJ. Cerebrovenous oxygen saturation monitoring: practical considerations and clinical relevance. Intensive Care Med. 2000 Aug;26(8):1028-36. doi: 10.1007/s001340051315. PMID 11030158
- [Background] Bailey DM, Taudorf S, Berg RM, Lundby C, McEneny J, Young IS, Evans KA, James PE, Shore A, Hullin DA, McCord JM, Pedersen BK, Moller K. Increased cerebral output of free radicals during hypoxia: implications for acute mountain sickness? Am J Physiol Regul Integr Comp Physiol. 2009 Nov;297(5):R1283-92. doi: 10.1152/ajpregu.00366.2009. Epub 2009 Sep 2. PMID 19726713